CLINICAL TRIAL: NCT05711381
Title: An Open-label, Single-dose Study to Evaluate the Pharmacokinetics, Safety and Tolerability of HM15912(Sonefpeglutide) in Subjects With Renal Impairment and Matched Control Subjects With Normal Renal Function
Brief Title: Phase 1 Study of PK and Safety of HM15912 (Sonefpeglutide) in Subjects With Normal and Severe Kidney Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HM-GLP2-102
Record Dates: First submitted 2022-11-08; First posted 2023-02-03 (Actual); Results first posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Renal Impairment
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Severe renal impairment (Experimental): Subjects with eGFR < 30mL/min/1.73m^2, but not requiring hemodialysis
  Interventions: Drug: HM15912
- Normal renal function (Experimental): Subjects with eGFR ≥ 90 mL/min/1.73m^2
  Interventions: Drug: HM15912
- Moderate renal impairment (Experimental): Subjects with 30 mL/min/1.73m^2 ≤ eGFR < 60 mL/min/1.73m^2
  Interventions: Drug: HM15912
- Mild renal impairment (Experimental): Subjects with 60 mL/min/1.73m^2 ≤ eGFR < 90 mL/min/1.73m^2
  Interventions: Drug: HM15912

INTERVENTIONS:
Drug: HM15912 — Singe subcutaneous administration of HM15912 0.5 mg/kg
  Other Names: Sonefpeglutide

SUMMARY:
An Open-label, Single-dose Study to Evaluate the Pharmacokinetics, Safety and Tolerability of HM15912 in Subjects with Renal Impairment and Matched Control Subjects with Normal Renal Function

DETAILED DESCRIPTION:
A single-dose, open-label, Phase 1 study (HM-GLP2-102) was conducted to evaluate the impact of renal impairment (RI) on the pharmacokinetics (PK) of HM15912. This study aimed to assess the safety and PK profile of HM15912 at a minimum effective dose of 0.5 mg/kg, which was determined based on findings from a previous clinical study (HM-GLP2-101).

The study was initially designed to be conducted in two parts.

Part 1: An open-label, single-dose, parallel-group study to investigate the effect of RI on the PK, safety, and tolerability of HM15912 in subjects with severe RI and subjects with normal renal function as a control group.

Part 2 (if applicable): An open-label, single-dose, parallel-group study to investigate the effect of RI on the PK, safety, and tolerability of HM15912 in subjects with moderate and mild RI.

ELIGIBILITY:
Inclusion Criteria:

All Subjects

* Subjects voluntarily agreed to participate in this study and sign an institutional review board (IRB)-approved informed consent form prior to performing any of the S1 procedures.
* Males and females ≥ 18 and ≤ 80 years of age at S1.
* Body mass index (BMI) of ≥ 17.5 to ≤ 40.0 kg/m^2.

Subjects with Normal Renal Function

* No clinically relevant abnormalities identified by detailed medical history, full physical examination, including blood pressure (BP) and heart rate (HR) measurements, 12-lead ECG, and clinical laboratory tests.
* Normal renal function (eGFR ≥ 90 mL/min/1.73m^2) at screening based on the chronic kidney disease-epidemiology collaboration (CKD-EPI) equation.
* Demographically comparable to the group of subjects with impaired renal function.

Subjects with Impaired Renal Function

* Met the following eGFR criteria during the screening period based on the CKD-EPI equation:

  1. Severe renal impairment: eGFR < 30 mL/min/1.73m^2, but not requiring hemodialysis.
  2. Moderate renal impairment: 30 mL/min/1.73m^2 ≤ eGFR < 60 mL/min/1.73m^2
  3. Mild renal impairment: 60 mL/min/1.73m^2 ≤ eGFR < 90 mL/min/1.73m^2

Exclusion Criteria:

All Subjects:

* Renal transplant recipients or subjects requiring hemodialysis and peritoneal dialysis.
* Subject with a history or presence of any psychiatric disorder that, in the opinion of the Investigator, might have confounded the results of the study or posed additional risk in administering the IP to the subject.
* Had participated in an interventional clinical trial (investigational or marketed product) within 1 month of screening or 5 half-lives of the drug under investigation (whichever came first), or planned to participate in another clinical trial.
* Subject with a history of any SAEs, hypersensitivity reactions, or intolerance to IP components.

Additional Exclusion Criteria for Subjects with Normal Renal Function

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal (GI), cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding treatment not required, asymptomatic, seasonal allergies at the time of dosing).
* Subject who had a mean BP ≥ 140 mmHg (systolic) or ≥ 90 mmHg (diastolic). After at least 5 minutes of supine rest, measurements were taken 2 consecutive times at least 2 minutes apart. If the mean of the 2 BP was ≥ 140mmHg (systolic) or ≥ 90 mmHg (diastolic), the BP should have been repeated 1 more time and the average of the 3 BP values should have been used to determine the subject's eligibility.
* Subject who had a baseline corrected QT using the Fridericia correction formula (QTcF) > 450 msec in males or QTcF > 470 msec in females.

Additional Exclusion Criteria for Subjects with Impaired Renal Function

* Subject with clinically significant active diseases that may have affected the safety of the subject or that may have affected the PK of HM15912 (including drug allergies, but excluding treatment not required, asymptomatic, seasonal allergies at time of dosing). Subjects with any significant hepatic, cardiac, or pulmonary disease or subjects who were clinically nephrotic. Hypertension, diabetes mellitus, hyperparathyroidism, ischemic heart disease, etc. were not causes for exclusion as long as the subject was medically stable and any drugs that were administered for these conditions were not expected to interfere with the PK of HM15912.
* Subject who had a mean BP ≥ 180 mm Hg (systolic) or ≥ 120 mm Hg (diastolic). After at least 5 minutes of supine rest, measurements were taken 2 consecutive times at least 2 minutes apart. If the mean of the 2 BP was ≥ 180 mm Hg (systolic) or ≥ 120 mmHg (diastolic), the BP should have been repeated 1 more time and the average of the 3 BP values should have been used to determine the subject's eligibility.
* Subject who had a baseline QTcF > 480 msec.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2022-12-02 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-08-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Orange County Research Center, Tustin, California
  - Clinical Pharmacology of Miami, Miami, Florida
  - Panax Clinical Research, Miami Lakes, Florida
  - AMR Knoxville, Knoxville, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A single-dose, open-label, phase 1 study, which was to characterize the effect of RI on the PK of HM15912, was planned to be conducted in 2 parts.
  A total of 16 subjects, 8 subjects with severe RI (Cohort 2) and 8 subjects with normal renal function (Cohort 1), were enrolled for Part 1.
  Part 2 of the study, which was optional to evaluate the effect of moderate and mild renal impairment on the PK of HM15912 following a single SC dose, was not conducted based on the results from Part 1.
Groups:
- Severe Renal Impairment: Subjects with eGFR < 30mL/min/1.73m^2, but not requiring hemodialysis, received 0.5 mg/kg SC dose of HM15912 on Day 1.
- Normal Renal Function: Subjects with eGFR ≥ 90 mL/min/1.73m^2, received 0.5 mg/kg SC dose of HM15912 on Day 1.
- Moderate Renal Impairment (Part 2 Only): Subjects with 30 mL/min/1.73m^2 ≤ eGFR < 60 mL/min/1.73m^2
- Mild Renal Impairment (Part 2 Only): Subjects with 60 mL/min/1.73m^2 ≤ eGFR < 90 mL/min/1.73m^2
Period: Overall Study
Arm/Group | Severe Renal Impairment | Normal Renal Function | Moderate Renal Impairment (Part 2 Only) | Mild Renal Impairment (Part 2 Only)
Started | 8 | 8 | 0 | 0
Completed | 8 | 8 | 0 | 0
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants
Groups:
- Severe Renal Impairment: Subjects with eGFR < 30 mL/min/1.73m^2, but not requiring hemodialysis, received 0.5 mg/kg SC dose of HM15912 on Day 1.
- Normal Renal Function: Subjects with eGFR≥ 90 mL/min/1.73m^2 received 0.5 mg/kg SC dose of HM15912 on Day 1.
- Total: Total of all reporting groups
Arm/Group | Severe Renal Impairment | Normal Renal Function | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Categorical [Count of Participants; unit: Participants] — Population: Safety population
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 4 | 8 | 12
    >=65 years | 4 | 0 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.3 (8.35) | 59.6 (3.25) | 61.4 (6.40)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Safety population
  Participants
    Female | 2 | 2 | 4
    Male | 6 | 6 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Safety population
  Participants
    Hispanic or Latino | 4 | 6 | 10
    Not Hispanic or Latino | 4 | 2 | 6
    Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8 | 8 | 16
Estimated glomerular filtration rate [Mean (Standard Deviation); unit: mL/min/1.73m^2] | 17.145 (7.5206) | 97.864 (4.2156) | 57.504 (42.0970)

OUTCOME MEASURES:

1. Primary Outcome: Maximum Serum Concentration (Cmax) of HM15912
Description: Pharmacokinetic (PK) samples were collected for measurement of serum concentrations of HM15912 and analyzed using a fully validated method.
Time Frame: Day 1 to 29 (Total duration: 29 days)
Population: PK population: All subjects who had at least one evaluable HM15912 serum concentration after receiving any amount of HM15912 without IPDs or events.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Severe Renal Impairment | Normal Renal Function
Number analyzed (Participants) | 8 | 8
ng/mL | 2811.25 (1498.985) | 3000.00 (1174.114)
Statistical Analysis 1: Comparison: Severe Renal Impairment vs Normal Renal Function; Test type: Other — PK parameters of HM15912 from the severe renal impairment group (Cohort 2) were to be estimated and compared to the control group (Cohort 1, normal renal function). A one-way analysis of variance (ANOVA) was to be used to compare log transformed PK parameters. The estimates of mean difference and corresponding 90% CIs, as well as each exponentiation of estimates, were to be presented to provide the estimates of GMR; Geometric mean ratio = 0.91, 90% CI 2-sided [0.59 to 1.41]

2. Primary Outcome: Area Under the Concentration-time Curve From Extrapolated to Infinity (AUC 0-infinity) of HM15912
Description: PK samples were collected for measurement of serum concentrations of HM15912 and analyzed using a fully validated method.
Time Frame: Day 1 to 29 (Total duration: 29 days)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Severe Renal Impairment | Normal Renal Function
Number analyzed (Participants) | 8 | 8
h*ng/mL | 1117469.3 (347572.67) | 890343.8 (235565.36)
Statistical Analysis 1: Comparison: Severe Renal Impairment vs Normal Renal Function; Test type: Other — [test comment as in outcome 1, analysis 1]; Geometric mean ratio = 1.25, 90% CI 2-sided [0.93 to 1.68]

3. Secondary Outcome: Overall Summary of Treatment-emergent Adverse Events (TEAEs)
Description: The number and percentages of subjects with TEAEs were to be summarized by cohort. A TEAE was defined as any AE that began, or worsened in severity, on or after the date of the first IP administration until the last follow-up visit.
Time Frame: Day 1 up to Day 29
Population: Safety Population: All subjects who received any amount of HM15912.
Measure: Count of Participants; unit: Participants
Arm/Group | Severe Renal Impairment | Normal Renal Function
Number analyzed (Participants) | 8 | 8
Participants
  Any Treatment-Emergent Adverse Events (TEAEs) | 1 | 1
  Any Treatment-Related Adverse Events (TRAEs) | 0 | 0
  Any Treatment-Emergent Serious Adverse Events (TESAEs) | 0 | 0
  Any TEAEs leading to Drug Interruption/Withdrawn | 0 | 0
  any TEAEs Leading to Death | 0 | 0

ADVERSE EVENTS:
Time Frame: From the signing of ICF util follow-up visit (about 2 months)
Description: Adverse Event (AE) analyses were to focus on Treatment-Emergent AEs (TEAEs), which were defined as any AE that began or worsened in severity on or after the date of the first IP administration until the last follow-up visit.
Arm/Group | Severe Renal Impairment | Normal Renal Function
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 1/8 | 1/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Severe Renal Impairment (N=8) | Normal Renal Function (N=8)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-08-05): https://cdn.clinicaltrials.gov/large-docs/81/NCT05711381/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-05): https://cdn.clinicaltrials.gov/large-docs/81/NCT05711381/SAP_001.pdf